CLINICAL TRIAL: NCT01710163
Title: ARIQUELI: Potentiation of Quetiapine Treatment in Bipolar 1 Nonresponders Patients With Lithium or Aripiprazole
Brief Title: Potentiation of Quetiapine Treatment With Lithium or Aripiprazole in Bipolar 1 Nonresponders Patients
Acronym: ARIQUELI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Alberto Moreno, M.D., Ph.D., MD PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARIQUELI
Record Dates: First submitted 2012-07-28; First posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Bipolar I Disorder
Keywords: Lithium Carbonate; Lithium; Central Nervous System Agents; Therapeutic Uses; Pharmacologic Actions; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Neurotransmitter Agents; Physiological Effects of Drugs; Antimanic Agents; Tranquilizing Agents; Central Nervous System Depressants; Psychotropic Drugs; Sensory System Agents; Antipsychotic Agents; Antidepressive Agents
MeSH Terms: interventions — Lithium; Aripiprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lithium (Experimental): Potentiation of previous treatment (Quetiapine monotherapy) with Lithium (0.5 - 0.8 mEq/L)
  Interventions: Drug: Lithium
- Aripiprazole (Experimental): Potentiation of previous treatment (Quetiapine monotherapy) with Aripiprazole (10 - 15 mg)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Lithium — Starting at 300 mg daily, weekly dose will be adjusted according to blood serum level (between 0.5 -0.8mEq/l) according to efficacy and tolerability.
  Arms: Lithium
Drug: Aripiprazole — Starting at 10 mg daily, dose will be adjusted up to 15 mg daily according to efficacy and tolerability.
  Arms: Aripiprazole

SUMMARY:
The purpose of this study is to determine whether Bipolar I Disorder refractory treatment with Quetiapine monotherapy could be better potentiated with Lithium or Aripiprazole. The investigators hypothesized that Lithium or Aripiprazole would provide similar compliance and tolerability in maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Bipolar Disorder, type I, in current episode (manic/hypomanic, mixed or depression)
* The patient or his (her) legal representative should understand the nature of the study and sign the Informed Consent

Exclusion Criteria:

* Schizophrenia or schizoaffective disorder
* Mental retardation
* Unstable clinical diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The main outcome will be the number of patients that achieve and remain in remission to each treatment at the end of each phase of the study | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Alberto Moreno, MD, PhD, Principal Investigator — Institute of Psychiatry, University of São Paulo; Giovani Missio, MD, Study Chair — Institute of Psychiatry, University of São Paulo
Locations (2):
- Brazil (2):
  - Institute of Psychiatry, University of São Paulo, São Paulo, São Paulo
  - Institute of Psychiatry, São Paulo, São Paulo

REFERENCES:
- [Derived] Missio G, Moreno DH, Fernandes F, Bio DS, Soeiro-de-Souza MG, Rodrigues dos Santos D Jr, David DP, Costa LF, Demetrio FN, Moreno RA. The ARIQUELI study: potentiation of quetiapine in bipolar I nonresponders with lithium versus aripiprazole. Trials. 2013 Jun 27;14:190. doi: 10.1186/1745-6215-14-190. PMID 23805994